CLINICAL TRIAL: NCT06045572
Title: Vascular Supply Identification, Lesion Extension and Search for Tumor Similarity at a Distance by VTM in Breast Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Galzu Institute of Research, Teaching, Science and Applied Technology (Other)
Collaborators: Hospital Santa Casa de Misericordia de Campos (Unknown); Hospital Escola Alvaro Alvim (Unknown); Universidade Estadual do Norte Fluminense (UENF) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IGZ-03
Record Dates: First submitted 2023-09-06; First posted 2023-09-21 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer Female

STUDY DESIGN:
Intervention Model Description: Pivotal, prospective, controlled study (comparison with genetic tests, histopathological / immunohistochemical analysis) to evaluate the safety and performance of VTM as a diagnostic test in breast cancer.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- women diagnosed with breast cancer before cancer treatment (Experimental)
  Interventions: Device: VTM examination and breast biopsy

INTERVENTIONS:
Device: VTM examination and breast biopsy — VTM examination performed by a radiologist, at the MART (Metabolic Activity in Real-Time) station, using the SaMD Mart 2.0, according to the inspection protocol to identify breast alterations and/or suspicious images to be biopsied for validation by genetic tests and histology / immunohistochemistry.

SUMMARY:
When we talk about early identification, we are talking about an ALREADY EXISTING INJURY, triggering a change in the patient's quality of life and a projection of future costs for the health system.

INNOVATIVE ASPECT: While screening mammography identifies an existing lesion, VTM could: Make an early diagnosis before the formation of a visible or palpable tumor mass; Check the metabolic activity in suspicious lesions identified by other diagnostic methods; Demarcate tumor range and tumor similarity from a distance in breast cancer.

Regarding the Risk x Benefit:There are no medications incorporated, associated or administered by the equipment; There is no ionizing radiation incorporated or delivered by the equipment; There are no contraindications for the use of the equipment by the patient (Non-ionizing infrared radiation, without contrast or contact); Audience destined to operate the equipment: Physician / Radiologist with training Therefore, the research in question is of great relevance for such a debilitating health problem for the patient and for the health system.

DETAILED DESCRIPTION:
Breast cancer control has been one of the priorities on the agenda of the National Health Policy in Brazil. Thus, the Ministry of Health, through the publication "Guidelines for the Early Detection of Breast Cancer in Brazil", recommends the identification of the disease in its early stages through early detection strategies. It is estimated that there will be 66,280 new cases of breast cancer for each year of the three-year period 2020-2022 in Brazil and Population-Based Cancer Registries (RCBP), Hospital Cancer Registries (RHC) and information on Mortality are essential requirements for national and regional programs for cancer control, in addition to guiding the research agenda.

According to the National Cancer Institute (INCA), the benefit of screening mammography is in early identification, allowing for less aggressive treatment.

VTM is a functional method that demonstrates the metabolic intensity in real time, through images in the colors of the visible spectrum without using ionizing energy or contrast. It expresses metabolic alterations before anatomical transformations. It is a method without radiation, contrast, pain or contact, and can be used without limiting the exposure time.

ELIGIBILITY:
Inclusion Criteria:

Women ≥18 years old; Women with breast cancer before oncological treatment; Voluntary signature of the Free and Informed Consent Term.

Exclusion Criteria:

Pregnant or lactating women; Patients already included in other clinical trials; Patients who are undergoing radiotherapy, chemotherapy or post-cancer surgery treatment; Patients who need urgent or emergency care; Patients with fever or other illness that affects the integrity of the skin; Any clinically significant medical condition or medical history that, in the opinion of the investigator, may discourage participation in the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-06-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Concordance of the diagnosis of abnormality during the VTM exam in relation to the standard exam (mammography); | [D2, approximately 60 days]
  Identification of the lesion (Yes/No); Identification of vascular alterations (Yes/No).
Frequency of non-visible vascular identification: | [D2, approximately 60 days]
  Vascular imaging (Yes/No); Vascular asymmetry (Yes/No); Thermal signature / tumor coverage (Yes/No). Identification of vascular alterations (Yes/No).
Frequency of identifying non-visible textures | [D2, approximately 60 days]
  Yes/No
Frequency of thermal discrepancy in nearby pixels in areas suspected of non-visible abnormalities: | [D2, approximately 60 days]
  Numerical (1 to 10)
Frequency of sample changes detected by VTM | [D2, approximately 60 days]
  Neoplastic, non-neoplastic and without alterations; Aggressiveness (Yes/No); Invasiveness (Yes/No); Presence of mutation (Yes/No); Gene expression: BRCA1/BRCA2, TP53, ATM, PTEN, STK11/LKB1 (Yes/No); Gene expression: S100P, NUP88 (2x, 3x, higher); Gene expression: ATP6V1C1 and TP6V1C2 (predominance of the C1/C2 isoform).

SECONDARY OUTCOMES:
(ClinROs) Diagnostic image quality by VTM in pathological changes of the breast; | [D2, approximately 60 days]
  Imaging data will be rated using a Likert scale by the study evaluator/radiologists (unacceptable, poor, acceptable, good, excellent);
(ClinROs) Ease of use and functionality; | [D2, approximately 60 days]
  easy/moderate/complex
(ClinROs) Image acquisition time; | [D2, approximately 60 days]
  fast/acceptable/long
(PROs) Discomfort during the VTM exam; | [D2, approximately 60 days]
  Y/N
(PROs) Pain during VTM exam; | [D2, approximately 60 days]
  Y/N
(PROs) Importance of the VTM exam research to the participant; | [D2, approximately 60 days]
  important/indifferent
Frequency of adverse events, unexpected adverse events, and serious adverse events (discrete numerical and categorical yes/no); | [D2, approximately 60 days]
  discrete numerical and categorical Y/N
All-cause mortality rate during the study; | [D2, approximately 60 days]
  numerical, %
Tolerability of the VTM exam; | [D2, approximately 60 days]
  Calculation of adherence to treatment; Proportion of participants who withdrew consent; Proportion of participants who dropped out of treatment.
Demographic data analysis; | [D1, approximately 01 day]
  Gender (F/M), age (Years), weight (Kg), height (m);
Demographic data analysis; | [D1, approximately 01 day]
  Past pathological history; Hormonal activity: pregnancy, breastfeeding, menarche and puerperium; Anamnesis, health history and complaints.
Prospective data. | [D1, approximately 01 day]
  Density of breast tissue; the size of the lesion; Degree of aggressiveness; BI-RADS classification.

IPD SHARING:
Plan to Share IPD: No